CLINICAL TRIAL: NCT02252601
Title: An Evaluation of the High Frequency Digit Triplet Test as a Screening Tool for Early Detection of Hearing Loss in Individuals With Cystic Fibrosis
Brief Title: Evaluation of the High Frequency Digit Triplet Test in Cystic Fibrosis
Acronym: 3D-CF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); Heart of England NHS Trust (Other); Birmingham Women's and Children's NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 3D-CF; PB-PG-0213-30055 (Other Grant/Funding Number: NIHR PB-PG-0213-30055)
Record Dates: First submitted 2014-09-17; First posted 2014-09-30 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Cystic Fibrosis; Sensorineural Hearing Loss
Keywords: Cystic Fibrosis; Hearing Loss; High Frequency Digit Triplet Test
MeSH Terms: conditions — Cystic Fibrosis; Hearing Loss, Sensorineural; Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Well patients aged 11 and over (Experimental): Will have the HFDT test compared to the gold standard (the Pure tone Audiogram) as well as other tests that have previously been suggested as a screening test for ototoxicity.
  Interventions: Other: HFDT test; Other: Pure tone Audiogram
- Acute exacerbation aged 11 and over (Experimental): Will have the HFDT test compared to the gold standard (the Pure tone Audiogram) as well as other tests that have previously been suggested as a screening test for ototoxicity at the beginning of a course of IV antibiotics and at their convalescent clinic visit.
  Interventions: Other: HFDT test; Other: Pure tone Audiogram
- Children with CF aged 5-10 years (Experimental): Will have the HFDT test compared to the gold standard (the Pure tone Audiogram) as well as other tests that have previously been suggested as a screening test for ototoxicity.
  Interventions: Other: HFDT test; Other: Pure tone Audiogram
- Healthy Control Children age 5-10 years. (Active Comparator): Will have the HFDT test compared to the gold standard (the Pure tone Audiogram) as well as other tests that have previously been suggested as a screening test for ototoxicity.
  Interventions: Other: HFDT test; Other: Pure tone Audiogram

INTERVENTIONS:
Other: HFDT test
Other: Pure tone Audiogram

SUMMARY:
The purpose of this study is to find out whether the High Frequency Digit Triplet test can be used to screen patients with cystic fibrosis for hearing loss in conditions of health and pulmonary exacerbation. It is also designed to find out the youngest age at which a child can perform the test, the prevalence of hearing loss in a CF population and the prevalence of genetic mutations known to be associated with hearing loss in the same population.

DETAILED DESCRIPTION:
Patients will be identified from the clinic list of four Cystic Fibrosis centres (Nottingham University Hospitals NHS (National Health Service) Trust, adults and children, West Midlands Adult Cystic Fibrosis Centre and Birmingham Children's Hospital).

In the first work stream patients 11 years old and over will answer some hearing screening questions and an ear examination and tympanogram. They will then have the new test (the High Frequency Digit Triplet, HFDT, test), the standard tests (Pure tone audiogram (PTA) including high frequencies, Distortion Product Otoacoustic Emissions) and then repeat the new test to look for order effect. These will be compared to validate the HFDT as a screening tool for hearing loss.

In the second work stream the investigators are looking to see if the test is feasible when a patient is unwell and about to start a course of IV antibiotics. The patients will have the same tests as in work stream 1 (though the high-frequency PTA may be modified if they are too unwell to complete it). They will then have the tests repeated at the next clinic visit (approximately 6-8 weeks later).

In the third work stream children aged 5-10 years will have the same tests. This is to discover the youngest age at which the HFDT test can reliably be performed. To ensure that the CF condition does not itself affect the ability to perform the test the investigators will compare CF children to healthy control children the same age.

The investigators will take blood and saliva samples from CF patients to look for mutations in mitochondrial genes which are known to be associated with aminoglycoside induced hearing loss.

ELIGIBILITY:
Inclusion criteria

Work stream 1

* A diagnosis of CF, confirmed by genotype or sweat test, with characteristic clinical features.
* Aged 11 years and over.
* Informed consent. For age 11 to 18 years, consent will be sought from both the parent and young person (provided the young person is competent).

Work stream 2

• As above but the participant has a pulmonary exacerbation (as defined by Fuch's criteria) requiring intravenous antibiotics.

Work stream 3

* As for work stream 1, defined above.
* CF patients aged 5-10 years
* Healthy control children aged 5-10 years.
* Informed consent from parent with assent from the child.

Genetic Testing

* Informed consent
* Diagnosis of CF as above

Exclusion criteria

* None. In individuals with a hearing aid, we will perform PTA and HFDT tests without the aid.
* Individuals found to have conductive deafness after randomisation will be fully assessed for this prior to continuing with the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in whom the HFDT test accurately predicts the presence of absence of hearing loss. | 2 years
  This will be done in patients when they are clinically stable and at the beginning and end of a pulmonary exacerbation by comparing the HFDT test with the current gold standard test.
The youngest age at which 80% of children are able to perform the HFDT test. | 2 years
  This will be done in children aged 5-10 years and the

SECONDARY OUTCOMES:
The prevalence of hearing loss in a CF population. | 2 years
The prevalence of genetic mutations that are associated with hearing loss in a CF population. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alan Smyth, MD, Principal Investigator — The University of Nottingham
Locations (3):
- United Kingdom (3):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Heart of England NHS Foundation Trust, Birmingham
  - Nottingham University Hospitals NHS Trust, Nottingham